CLINICAL TRIAL: NCT05980741
Title: Exploration of New Nursing Models for Urological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YaNi Peng (Other)
Responsible Party: Sponsor-Investigator, YaNi Peng, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TJ-IRB20220940
Record Dates: First submitted 2023-07-19; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Urological Nursing
Keywords: High-quality nursing, Primary nursing, Roy Adaptation Model, Urological surgery
MeSH Terms: interventions — Primary Nursing

STUDY DESIGN:
Intervention Model Description: High-quality nursing will be provided to the study group based on primary nursing
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): Traditional nursing services are provided to the control group, based on functional nursing. The nurses in the ward are assigned to complete different tasks according to their responsibilities, technical knowledge and skills. These tasks are including carrying out health education to the patients, introducing the admission guidelines and ward conditions, informing patients of basic knowledge on diseases, treatment, and nursing, monitoring patient vital signs and so on. The basic medical inspection and care are conducted appropriately. The patients are instructed on the compliance and precautions required during the perioperative period. The wound and drainage are checked regularly after the operation.
- study group High-quality nursing (Experimental): High-quality nursing is provided to the study group based on primary nursing. Nurses in primary nursing take responsibility for the total care of a patient and are accountable for his/her care over 24 h a day from the patient's admission to discharge. In this case, nurses have more time to communicate with patients and to establish the nurse-patient relationship. In addition, high-quality nursing offers effective nursing measures to patients in terms of multiple aspects and dimensions through planning patient-centered nursing care, strengthening the perioperative nursing since admission, and fully implementing the nursing responsibility system.
  Interventions: Procedure: high-quality nursing
- study group Clinical Care Pathway (Experimental): The clinical care pathway will be implemented immediately after admission. With the patient as the center of the nursing intervention, a flowable form is chosen to ensure that patients could receive effective nursing interventions throughout the entire hospitalization from the day of admission to the final discharge. In addition to primary care, the present program also unifies the management of nursing resources with the establishment of a highly qualified and professionally competent nursing team. The team members would cooperate with each other and give full play to their respective initiatives, with the common goal of improving the quality of care. The severity of illness, psychological status, and family and social environment in each patient differ, so individualized care plans are developed for each case.
  Interventions: Procedure: Clinical Care Pathway
- study group Roy Adaptation Model (Experimental): the Roy Adaptation Model (RAM) offers a comprehensive framework to guide nursing care for patients with chronic diseases. The RAM group receives standard care supplemented with interventions based on the RAM model. Negative emotions measured by the Hospital Anxiety and Depression Scale (HADS), pain intensity by the Visual Analog Scale (VAS), and HRQoL by the 36-Item Short Form Health Survey (SF-36) are measured at the preoperative visit (T0), at 30 days (T1), and at 3 months of (T2) follow-up.
  Interventions: Procedure: Roy Adaptation Model

INTERVENTIONS:
Procedure: high-quality nursing — High-quality nursing
  Other Names: primary nursing
  Arms: study group High-quality nursing
Procedure: Clinical Care Pathway — Clinical Care Pathway
  Arms: study group Clinical Care Pathway
Procedure: Roy Adaptation Model — Roy Adaptation Model
  Arms: study group Roy Adaptation Model

SUMMARY:
Patients undergoing urological surgery often need to be provided with targeted nursing care to ensure that the therapeutic effects can be fully realized, however, the traditional nursing cannot reach the expect effect.both patient outcome and nurse satisfaction have been reported with high levels of dissatisfaction in the traditional nursing. Therefore, exploring a new, patient-centered and effective nursing mode is needed. In 2010, the Chinese Ministry of Health proposed a project named the High-Quality Care Project to improve nurse and patient outcomes through the transformation of the nursing care delivery system in hospitals. This study aims to compare the new nursing model and the traditional nursing, and to explore a more effective nursing model for urological surgery.

DETAILED DESCRIPTION:
Patients who underwent urological disease diagnosed and treated in our department were included in this study. The patients were randomly divided into two groups through the random number table method, with a 1:1 ratio. The control group received traditional urological care. The study group comprised 3 subgroups, and each subgroup received different nursing model. All the three new nursing models, including high-quality nursing (primary nursing), Clinical care pathway, and Roy adaptation model.were given to the subgroups respectively.

High-quality nursing refers to effective nursing measures in multiple aspects and dimensions, provided to patients according to their actual conditions by centering on the patients throughout their ongoing treatment, strengthening the primary nursing care, and fully implementing the nursing responsibility including managing complications and providing long-term support and information, to ensure patient satisfaction and to improve the patient's quality of life. Clinical care pathway includes multidisciplinary care plans that provides detailed guidelines for patients with specific clinical problems, and the Roy adaptation model (RAM), proposed by nursing scientist Sister Callista Roy in 1970, offers a comprehensive framework to guide nursing care for patients with chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a definite diagnosis of urological disease confirmed by pathological examination or imaging;
2. patients with definite surgical indications;
3. patients with complete follow-up information.

Exclusion Criteria:

1. patients with hepatic or renal dysfunction or serious organic lesions in other organs;
2. patients with associated lymph node and distant metastases;
3. patients who withdrew during the study;
4. patients with incomplete case and follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Patients' quality of life after surgery | 3 months
  the 36-Item Short Form Health Survey (SF-36)
Patient satisfaction | 3 months
  The patient satisfaction was evaluated by means of an adapted version of Press-Ganey PS scores, which included physician-specific questions and hospital performance questions
Postoperative complications | 3 months
  Postoperative complications include hemorrhage, infection, and anuria
The postoperative time to flatus | 1 month
  postoperative recovery 1
the time for first bowel movement | 1 month
  postoperative recovery 2
the length of hospital stay | 1 month
  postoperative recovery 3

CONTACTS AND LOCATIONS:
Overall Officials: E-Jun Peng, Dr., Principal Investigator — Tong Ji Hospital, Tong Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No